CLINICAL TRIAL: NCT04137614
Title: The Effects and Safety of Drug-coated Balloon in the Treatment of Hypertension Caused by Takayasu Arteritis Associated Renal Artery Stenosis: a Single Centre, Random, Double Blind Trial
Brief Title: Drug-coated Balloon for Takayasu Arteritis Associated Renal Artery Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Jiang lindi, Shanghai Zhongshan Hospital, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TADCB2019
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Takayasu Arteritis
MeSH Terms: conditions — Takayasu Arteritis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital substraction angiography (Placebo Comparator)
  Interventions: Procedure: Digital substraction angiography (DSA)
- Drug-coated balloon (Experimental)
  Interventions: Procedure: Drug coated balloon (DCB)

INTERVENTIONS:
Procedure: Drug coated balloon (DCB) — Drug coated balloon (DCB）is a new type of PTA, which could improve the re-stenosis rate significantly.
  Arms: Drug-coated balloon
Procedure: Digital substraction angiography (DSA) — DSA was used to evaluated the stenosis of renal artery
  Arms: Digital substraction angiography

SUMMARY:
Takayasu arteritis associated renal artery stenosis (TARAS) is the biggest cause of hypertension in young people <40 years old. Hypertension caused by renal artery stenosis is usually hard to control in spite of two or more anti-hypertension drugs.

Percutaneous transluminal angioplasty (PTA) is recommended for hypertension caused by TARAS. In previous clinical practice, we observed relatively effects of PTA on controlling the blood pressure in patients with TARAS. But, high re-stenosis rate was also indicated. Drug coated balloon (DCB）is a new type of PTA, which could improve the re-stenosis rate significantly. In the clinical trials of peripheral vascular disease, it has been confirmed that DCB had lower re-stenosis rate than PTA. However, up to date, no studies was found about the use of DBC in TARAS.

Thus, this study was design as a random, double blind trial to evaluated the effects and safety of DCB in the treatment of hypertension caused by TARAS.

ELIGIBILITY:
Inclusion Criteria:

1. 18-60 years old;
2. diagnosed as Takayasu arteritis according to 1990 ACR classification
3. renal artery stenosis is confirmed by imaging results
4. had inactive disease, and the dose of glucocorticoids <10mg/day
5. blood pressure >160/90mmHg in spite of two or more antihypertensive drug
6. had no surgery of renal artery, including PTA, stent, or others.

Exclusion Criteria:

1. blood pressure >200/120mmHg in spite of two or more antihypertensive drug
2. had severe disease conditions
3. allergy to contrast agent
4. had other autoimmune disease
5. had severe abnormal lab test result

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-30 (Actual); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
the control of blood pressure after DCB | 6 month

SECONDARY OUTCOMES:
the re-stenosis rate after DCB | 6 month
the control of blood pressure after DCB | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Lindi Jiang, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Maksimowicz-McKinnon K, Clark TM, Hoffman GS. Limitations of therapy and a guarded prognosis in an American cohort of Takayasu arteritis patients. Arthritis Rheum. 2007 Mar;56(3):1000-9. doi: 10.1002/art.22404. PMID 17328078
- [Background] Misra DP, Wakhlu A, Agarwal V, Danda D. Recent advances in the management of Takayasu arteritis. Int J Rheum Dis. 2019 Jan;22 Suppl 1:60-68. doi: 10.1111/1756-185X.13285. PMID 30698358
- [Background] Ishikawa K, Maetani S. Long-term outcome for 120 Japanese patients with Takayasu's disease. Clinical and statistical analyses of related prognostic factors. Circulation. 1994 Oct;90(4):1855-60. doi: 10.1161/01.cir.90.4.1855. PMID 7923672
- [Result] van den Berg JC. Drug-eluting balloons for treatment of SFA and popliteal disease - A review of current status. Eur J Radiol. 2017 Jun;91:106-115. doi: 10.1016/j.ejrad.2017.03.015. Epub 2017 Mar 27. PMID 28629556
- [Result] Schroe H, Holden AH, Goueffic Y, Jansen SJ, Peeters P, Keirse K, Ito W, Vermassen F, Micari A, Blessing E, Jaff MR, Zeller T. Stellarex drug-coated balloon for treatment of femoropopliteal arterial disease-The ILLUMENATE Global Study: 12-Month results from a prospective, multicenter, single-arm study. Catheter Cardiovasc Interv. 2018 Feb 15;91(3):497-504. doi: 10.1002/ccd.27348. Epub 2017 Oct 31. PMID 29086462
- [Result] Thieme M, Von Bilderling P, Paetzel C, Karnabatidis D, Perez Delgado J, Lichtenberg M; Lutonix Global SFA Registry Investigators. The 24-Month Results of the Lutonix Global SFA Registry: Worldwide Experience With Lutonix Drug-Coated Balloon. JACC Cardiovasc Interv. 2017 Aug 28;10(16):1682-1690. doi: 10.1016/j.jcin.2017.04.041. Epub 2017 Aug 2. PMID 28780030
- [Result] Micari A, Brodmann M, Keirse K, Peeters P, Tepe G, Frost M, Wang H, Zeller T; IN.PACT Global Study Investigators. Drug-Coated Balloon Treatment of Femoropopliteal Lesions for Patients With Intermittent Claudication and Ischemic Rest Pain: 2-Year Results From the IN.PACT Global Study. JACC Cardiovasc Interv. 2018 May 28;11(10):945-953. doi: 10.1016/j.jcin.2018.02.019. PMID 29798770
- [Result] Zhu G, He F, Gu Y, Yu H, Chen B, Hu Z, Liang W, Wang Z. Angioplasty for pediatric renovascular hypertension: a 13-year experience. Diagn Interv Radiol. 2014 May-Jun;20(3):285-92. doi: 10.5152/dir.2014.13208. PMID 24675165
- [Result] Kim YW, Sung K, Park YJ, Kim DK. Surgical treatment of middle aortic syndrome due to Takayasu arteritis. J Vasc Surg. 2015 Sep;62(3):750-1. doi: 10.1016/j.jvs.2014.05.017. No abstract available. PMID 26304483
- [Result] Kinjo H, Kafa A. The results of treatment in renal artery stenosis due to Takayasu disease: comparison between surgery, angioplasty, and stenting. A monocentrique retrospective study. G Chir. 2015 Jul-Aug;36(4):161-7. doi: 10.11138/gchir/2015.36.4.161. PMID 26712071